CLINICAL TRIAL: NCT05445037
Title: Hemodynamic and Cerebral Effect of General Anesthesia Plus Block Interescalenic vs Sedation Plus Block Interescalenic: The Recognised Randomized Controlled Trial
Brief Title: Hemodynamic and Cerebral Effects Evaluation in Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo (Other)
Responsible Party: Principal Investigator, João manoel Silva Junior, PhD, Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USP
Record Dates: First submitted 2022-06-01; First posted 2022-07-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hemodynamic Monitoring; Orthopedic Procedures

STUDY DESIGN:
Intervention Model Description: The selected patients will be divided into two groups: group 1 general anesthesia + interscalene brachial plexus block and group 2 sedation + interscalene brachial plexus block. Each group will be divided into two groups, one with hemodynamic continuous monitoring and one with standard hemodynamic monitoring, totaling 4 groups in total in the study. Group 1A general anesthesia + interscalene brachial plexus block with continuous monitoring; group 1B general anesthesia + interscalene brachial plexus block with standard monitoring; group 2A sedation + interscalene brachial plexus block with continuous monitoring; group 2B sedation + interscalene brachial plexus block with standard monitoring.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuos Monitoring (Experimental): Continuos monitoring will be done with clearsight continuously assessing blood pressure, cardiac output and heart rate; NIRS electrode to access cerebral O2 saturation, peripheral O2 saturation, BIS value and axillary temperature.
  Interventions: Device: hemodynamic continuous monitoring
- Standard monitoring (Experimental): Standard monitoring will be done with non-invasive
  Interventions: Device: Standard Monitoring

INTERVENTIONS:
Device: hemodynamic continuous monitoring — Continuous monitoring will be done with clearsight continuously assessing blood pressure, cardiac output and heart rate; NIRS electrode to assess cerebral O2 saturation, peripheral O2 saturation, BIS value and axillary temperature.
  Arms: Continuos Monitoring
Device: Standard Monitoring — Standard monitoring will be done with non-invasive blood pressure, heart rate, NIRS electrode to access cerebral O2 saturation, peripheral O2 saturation, axillary temperature, BIS value. In addition, patients will use Clearsight, but the device will be blind to the anesthesiologist. Pressure monitoring will be every 5 min.
  Arms: Standard monitoring

SUMMARY:
Recently, there has been an increase in the popularity of minimally invasive surgical techniques, including arthroscopic surgeries for shoulder procedures. Interscalene block is currently the gold standard technique for these surgeries, combined or not with general anesthesia. The last, when used in patients positioned in a beach chair can lead to serious hemodynamic and cerebral changes in the patients. Continuous non-invasive monitoring of the patient's cardiac output can provide data for better hemodynamics management compared to standard monitoring. Therefore, the aim of the study is to compare hemodynamic changes (cardiac output, blood pressure, heart rate, oxygen saturation) and intraoperative cerebral oxygenation using peripheral cerebral saturation monitoring with continuous measurement of cardiac output or standard hemodynamic between two anesthetic techniques for shoulder surgery: interscalene block with sedation versus interscalene block with general anesthesia. The groups will be evaluated as follows: group 1 general anesthesia plus interscalene brachial plexus block and group 2 sedation plus interscalene brachial plexus block. Additionally, each group will be subdivided into two more groups, one with continuous hemodynamic monitoring and the other with standard hemodynamic monitoring, that is, a total of 4 groups in the study. The analyzed variables will include gender, age, ASA, medications in use, comorbidities. Furthermore, duration of procedure and in the anesthetic recovery room, blood pressure, heart rate, cardiac output, peripheral oxygen saturation, cerebral oxygen saturation, BIS value, cardiac index, etCO2 will be evaluated. Besides, length of hospital stay, delirium, behavioral status and postoperative complication will also be assessed.

DETAILED DESCRIPTION:
The study will be split in 4 groups, being group 1A general anesthesia plus interscalene brachial plexus block with continuos non-invasive monitoring, group 1B general anesthesia plus interscalene brachial plexus block with standard hemodynamic monitoring, group 2A sedation plus interscalene brachial plexus block with continuos non-invasive monitoring, gruop 2B sedation plus interscalene brachial plexus block with standard hemodynamic monitoring.

The standard hemodynamic monitoring includes blood pressure, heart rate, peripheral oxygen saturation, brain monitoring and cerebral oxygen saturation. The continuos non-invasive monitoring includes the standard monitoring plus cardiac output, cardiac index and hypotension predict index. These variables will be analyzed intraoperatively and compared between groups with the aim of demonstrating the benefit of continuous non-invasive monitoring.

In the postoperative will be evalueted delirium, lenght hospital stay, postoperative complication and pain. We will use the Richmond Agitation Sedation Scale (RASS), Confusion Assessment Method in the ICU, visual analogue pain scale and visual numeric pain scale for evaluation postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing arthroscopic shoulder surgery in a beach chair position.

Exclusion Criteria:

* Emergency surgery
* Blood dyscrasia
* Refusal of the procedure
* Infection at the puncture site
* Allergy to the medication used
* Previous cerebrovascular disease
* History of orthostatic hypotension
* Pulmonary disease
* Chronic use of opioids
* Performance of arthroscopic surgeries on both shoulders
* Refusal to participate in the study
* Not to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-16 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Compare intraoperative hemodynamic changes: cardiac output | Intraoperative
  Compare cardiac output changes between continuous hemodynamic measurement of cardiac output or standard hemodynamics monitoring in two anesthetic techniques for shoulder surgery: interscalene block with sedation versus interscalene block with general anesthesia.
Compare intraoperative hemodynamic changes: blood pressure | Intraoperative
  Compare blood pressure changes between continuous hemodynamic measurement of cardiac output or standard hemodynamics monitoring in two anesthetic techniques for shoulder surgery: interscalene block with sedation versus interscalene block with general anesthesia.
Compare intraoperative hemodynamic changes: heart rate | Intraoperative
  Compare heart rate changes between continuous hemodynamic measurement of cardiac output or standard hemodynamics monitoring in two anesthetic techniques for shoulder surgery: interscalene block with sedation versus interscalene block with general anesthesia.
Evaluation of continuos hemodinamic monitoring non-invasive | Intraoperative
  Verify the superiority of continuos hemodynamic non-invasive monitoring of cardiac output compared to standard hemodynamic monitoring regarding blood pressure
Evaluation of cerebral tissue saturation | Intraoperative
  Compare changes in cerebral tissue saturation between groups

CONTACTS AND LOCATIONS:
Overall Officials: João M Silva Junior, PhD, Study Director — Instituto de Assistencia Medica ao Servidor Publico Estadual, Sao Paulo
Locations (1):
- Hospital do Servidor Público Estadual de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT05445037/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/37/NCT05445037/ICF_001.pdf